CLINICAL TRIAL: NCT04159285
Title: Augmenting and Sustaining Electroconvulsive Therapy (ECT) Treatment Effects by Group Cognitive Behavioural Therapy (CBT) in Unipolar Depressed Patients
Brief Title: Psychotherapeutic Augmentation of Brain Stimulation Effects
Acronym: PAUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Simone Grimm, Prof. Dr.rer.nat. Simone Grimm, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAUSE
Record Dates: First submitted 2019-08-01; First posted 2019-11-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Depression Chronic; Depression, Unipolar; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CBT (Experimental): 15-week group CBT with a focus on improvement of social interactions by cognitive re-modelling and role plays. Patients may simultaneously receive continuation ECT and/or individual psychotherapy and/or take anti-depressive medication.
  Interventions: Behavioral: EffEKTiv 2.0 group CBT as continuation treatment after ECT in depressed patients; Other: Treatment as usual
- Treatment as Usual (Experimental): Patients may receive continuation ECT and/or individual psychotherapy and/or take anti-depressive medication.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: EffEKTiv 2.0 group CBT as continuation treatment after ECT in depressed patients — Group CBT with a maximum number of 8 participants. Group is half-open allowing a starting date right after completion of acute ECT treatment. Patients participate for 15 sessions, which are framed by 2 individual sessions before joining the group and one individual session at treatment end.
  Arms: Group CBT
Other: Treatment as usual — Can include continuation ECT, psychopharmacological treatment, individual psychotherapy

SUMMARY:
This study aims to investigate effectiveness and feasability of a 15-week group psychotherapeutic intervention as continuation treatment after electroconvulsive therapy in severely depressed patients. Feasibility and acceptance of the half-open manualized CBT intervention are assessed. Depressive symptoms, quality of life and emotion regulation skills will be assessed before ECT treatment, before and after the 15-week group CBT intervention and at a 6 months follow-up after treatment end and compared to depressed patients treated with ECT who did not partake in group CBT. Moreover, patients will attend two indidivual pre-group sessions with one of the group therapist and one individual post-group session

DETAILED DESCRIPTION:
While Electroconvulsive therapy (ECT) is a highly effective anti-depressant treatment, a relevant number of patients experience recurrence of depressive episodes within 6 months.

One previous study suggested that ECT treatment effects can be effectively sustained by group CBT (Cognitive Behavioral Therapy, Brakemeier et a. 2014). This previous implementation used a closed CBT-group set-up that implicated a longer waiting period for patients after finishing the acute ECT and did not investigate whether patients who did not respond to ECT could sufficiently profit from group CBT. In order to suit the complex needs of patients in a natural clinical setting, the present study aims to investigate the feasibility and effectiveness of a half-open continuous group CBT (named EffECtive 2.0) as continuation treatment for all ECT patients regardless of remission status after ECT.

This prospective study will recruit a total of 30 patients who concluded treatment with right-unilateral ultra-brief ECT for depression. Patients self-allocate to the group that is offered in addition to continuation treatment as usual (TAU, e.g. pharmacological treatment, continuation ECT, individual psychotherapy). ECT completers who choose not to partake in the group for practical concerns or lack of interest and receive treatment as usual are recruited as a control group.

The primary outcome measure is the change depression severity, measured with the Montgomery-Åsberg Depression Rating Scale (MADRS). Secondary outcomes are quality of life assessed with the short-version of the WHO quality of life questionnaire (WHOQOL-Bref) and emotion regulation as assessed with cognitive emotion regulation questionnaire (CERQ). These measures will be assessed before, during, immediately after acute ECT and six and 12 months into continuation therapy.

It is hypothesized that a group CBT as add-on treatment to TAU will lead to more favorable outcomes concerning depression severity, quality of life and emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* treated with ECT for major depression

Exclusion Criteria:

* severe comorbid personality disorders
* principal diagnosis other than depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Clinican-Rated Depressive Symptoms at treatment end | End of group therapy treatment (~6 months after ECT treatment)
  MADRS
Clinican-Rated Depressive Symptoms at follow-up | 6 months after end of group therapy
  MADRS

SECONDARY OUTCOMES:
Quality of life at follow-up | 6 months after end of group therapy
  WHOQL-Bref
Emotion regulation capacities at follow-up | 6 months after end of group therapy
  Cognitive Emotion Regulation Questionnaire
Self-Reported Depressive Symptoms at treatment end | End of group therapy treatment (~6 months after ECT treatment)
  BDI
Self-Reported Depressive Symptoms at follow up | 6 months after end of group therapy
  BDI

CONTACTS AND LOCATIONS:
Overall Officials: Simone Grimm, Prof. Dr., Principal Investigator — Charite Universitaetsmedizin
Locations (1):
- Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brakemeier EL, Merkl A, Wilbertz G, Quante A, Regen F, Buhrsch N, van Hall F, Kischkel E, Danker-Hopfe H, Anghelescu I, Heuser I, Kathmann N, Bajbouj M. Cognitive-behavioral therapy as continuation treatment to sustain response after electroconvulsive therapy in depression: a randomized controlled trial. Biol Psychiatry. 2014 Aug 1;76(3):194-202. doi: 10.1016/j.biopsych.2013.11.030. Epub 2013 Dec 12. PMID 24462229